CLINICAL TRIAL: NCT02756975
Title: Prostate Core Needle Biopsy
Acronym: Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modarres Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Prostate Core Needle Biopsy
Record Dates: First submitted 2016-04-26; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Biopsy; Prostate; Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- transperineal prostate biopsy with coaxial method (Experimental): The patients undergo transperineal biopsy with a coaxial Tru-Cut needle (18-gauge Core Biopsy Instrument with a 17-gauge Disposable Coaxial Needle).
  Interventions: Device: coaxial prostate biopsy
- transperineal prostate biopsy with noncoaxial method (Experimental): The patients undergo transperineal biopsy with a noncoaxial 18-gauge needle.
  Interventions: Device: noncoaxial prostate biopsy

INTERVENTIONS:
Device: coaxial prostate biopsy — In this method, a larger introducing needle is needed for the puncture. The introducing needle is placed over the perineum. The biopsy needle is inserted throughout the introducing needle.Then, the direction of the biopsy is changed by tilting the coaxial needle. The investigator needs to puncture the prostate capsule only once for sampling at each each side of the prostate (right and left sides).
  Other Names: coaxial Tru-Cut needle (18-gauge Bard Max-Core Disposable Core Biopsy Instrument, 17-gauge Bard TruGuide Disposable Coaxial Needle; C. R. Bard, Tempe, USA)
  Arms: transperineal prostate biopsy with coaxial method
Device: noncoaxial prostate biopsy — In this method, there is no introducing needle. Biopsy needle is inserted repeatedly for each tissue sampling (at least fourteen times). A smaller biopsy needle is used for the puncture in this method.
  The main disadvantage of the coaxial technique is that a larger introducing needle is needed for the puncture (12). On the other whand, the advantage of noncoaxial method is that the needle is within the prostate for only a few seconds to document needle position with ultrasonography before firing
  Other Names: noncoaxial 18-gauge needle (Bard Max-Core Disposable Core Biopsy Instrument; C. R. Bard, Tempe, USA)
  Arms: transperineal prostate biopsy with noncoaxial method

SUMMARY:
Prostate tissue biopsy is performed with either transrectal or transperineal approach. These two methods are usually based on tissue sampling with an ultrasound-guided core needle biopsy. Transperineal prostate biopsy can be done either with a conventional noncoaxial technique or with a coaxial technique. In conventional transperineal technique, biopsy needle is inserted repeatedly for each tissue sampling. Alternatively, a coaxial needle can be placed over the perineum; then, the direction of the biopsy can be changed by tilting the coaxial needle. In this prospective study, the investigators sought to compare the procedural time and the complication rate of coaxial technique with those of noncoaxial technique in transperineal prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* an elevated prostate-specific antigen (PSA) level
* suspicious digital rectal examination

Exclusion Criteria:

* a history of prostate cancer
* clinical findings of acute or chronic prostate inflammation
* a history of urogenital procedures

Ages: 20 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
complication ratio | within 48 hours after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Poursina Hospital, Guilan University of Medical Sciences, Rasht, Gilan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Novella G, Ficarra V, Galfano A, Ballario R, Novara G, Cavalleri S, Artibani W. Pain assessment after original transperineal prostate biopsy using a coaxial needle. Urology. 2003 Oct;62(4):689-92. doi: 10.1016/s0090-4295(03)00483-7. PMID 14550444
- [Result] Chang DT, Challacombe B, Lawrentschuk N. Transperineal biopsy of the prostate--is this the future? Nat Rev Urol. 2013 Dec;10(12):690-702. doi: 10.1038/nrurol.2013.195. Epub 2013 Sep 24. PMID 24061531